CLINICAL TRIAL: NCT07108894
Title: A First-in-Human Phase 1 Single-Ascending Dose Study of ABCL575 in Healthy Participants
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: AbCellera Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABCL575-101; 297628 (Other: Health Canada CTA control number)
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABCL575 (Experimental): Healthy participants will receive a single dose of ABCL575 administered by subcutaneous (SC) injection
  Interventions: Biological: ABCL575
- Placebo (Placebo Comparator): Healthy participants will receive a single dose of placebo administered by subcutaneous (SC) injection
  Interventions: Biological: Placebo (Normal Saline 0.9%)

INTERVENTIONS:
Biological: ABCL575 — Participants will receive SC injection of ABCL575
  Arms: ABCL575
Biological: Placebo (Normal Saline 0.9%) — Participants will receive SC injection of placebo (Normal Saline 0.9%)
  Arms: Placebo

SUMMARY:
This study aims to assess the safety and tolerability of ABCL575 in healthy participants following single ascending dose (SAD), in comparison to a placebo

DETAILED DESCRIPTION:
This is a phase I randomized, double-blind, placebo-controlled, single ascending dose (SAD) study. The study will consist of 4 planned cohorts (A1 to A4), each comprised of 8 healthy participants. Doses of ABCL575 are intended to escalate through cohorts A1 to A4.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female ≥ 18 and ≤ 65 years of age at the time of screening
* Good general health as determined through medical history and general physical examination
* Body weight ≥ 50 and ≤ 100 Kg
* Body mass index (BMI) between 18.5 kg/m2 and 30.0 kg/m2
* Non- or ex-smoker (an ex-smoker defined as someone who has completely stopped using nicotine products for at least 180 days prior to study drug administration)
* Meeting 1 of the following:

  1. Is of childbearing potential or able to procreate and agrees to use an acceptable contraceptive method from at least 28 days prior to the screening visit through EOS visit
  2. Is of nonchildbearing potential or unable to procreate
* If male, agrees not to donate sperm from the study drug administration through EOS visit; If female, agrees not to donate or retrieve eggs from the study drug administration through EOS visit

Exclusion Criteria:

* Pregnancy and/or lactation.
* Seated pulse rate less than 50 beats per minute (bpm) or more than 100 bpm or a seated blood pressure < 90/50 mmHg or > 140/90 mmHg
* eGFR < 60 mL/min/1.73 m2
* Severe hypersensitivity reactions (like angioedema) to any drugs.
* Presence or history of significant gastrointestinal, liver disease, kidney disease, or surgery that may affect drug bioavailability.
* History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease.
* History or presence of multiple or severe drug allergies.
* Evidence of any active bacterial, viral, or fungal infection
* Disrupted skin integrity (apparent burn or dermatitis).
* History of syncope, palpitations, or unexplained dizziness.
* Use of prescription drugs (except for hormonal contraceptives or hormone replacement therapy) in the 28 days prior to study drug administration.
* Use of any over-the-counter products in the 7 days prior to study drug administration.
* Receipt of live vaccines within 5 weeks prior to screening or plans to receive live vaccines within 180 days after study drug administration.
* History of latent or active tuberculosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence, frequency, and severity of adverse events (AEs) | Day 0 to day 337
Changes from baseline in laboratory parameters including general biochemistry, lipid profile, coagulation, hematology, and urinalysis | Day 0 to day 337
Changes from baseline in physical examination | Day 0 to day 337
Changes from baseline in vital signs | Day 0 to day 337
Changes from baseline in 12-lead safety ECGs | Day 0 to day 337
Incidence and severity of injection site reactions | Day 0 to day 337

SECONDARY OUTCOMES:
Plasma concentrations of ABCL575 | Day 0 to day 337
Incidence of anti-ABCL575 antibodies | Day 0 to day 337
PK parameters; maximum plasma concentration (Cmax) | Day 0 to day 337
PK parameters; time to maximum plasma concentration (Tmax) | Day 0 to day 337
PK parameters; area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration (AUC0-T) | Day 0 to day 337
PK parameters; area under the plasma concentration-time curve from zero to hour 672 (AUC0-672) | Day 0 to day 337
PK parameters; area under the plasma concentration-time curve from zero to infinity (AUC0-∞) | Day 0 to day 337
PK parameters; terminal rate constant (λz) | Day 0 to day 337
PK parameters; apparent plasma clearance of drug after extravascular administration (CL/F) | Day 0 to day 337
PK parameters; apparent volume of distribution after extravascular administration (Vz/F) | Day 0 to day 337
PK parameters; half-life (Thalf) | Day 0 to day 337

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, Principal Investigator — Altasciences Company Inc.
Locations (1):
- Altasciences Company Inc., Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No